CLINICAL TRIAL: NCT00004639
Title: Velopharyngeal Function for Speech After Palatal Surgery
Brief Title: Cleft Palate Surgery and Speech Development
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDCR-010; R01DE010437 (NIH); NCT00004462 (obsolete NCT alias)
Record Dates: First submitted 1999-09-17; First posted 1999-09-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-06

CONDITIONS: Cleft Lip; Cleft Palate
Keywords: cleft lip and palate; children; speech; velopharyngeal function; congenital facial malformation; von Langenbeck procedure; Furlow procedure; cleft lip and palate repair; Unilateral cleft lip and palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Speech

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Furlow double z-plasty palatoplasty palate repair
Procedure: Von Langenbeck palatoplasty palate repair

SUMMARY:
Compare the outcome of two primary surgeries techniques (von Langenbeck and Furlow double z-plasty) performed on children with cleft lip/palate to determine if one results in significantly better velopharyngeal competency for speech.

DETAILED DESCRIPTION:
This study is conducted with patients with complete unilateral cleft lip and palate. The subjects will have their palatal clefts surgically repaired by either the von Langenbeck or the Furlow double z-plasty palatoplasty. Patients will be randomly assigned to four groups, to have with the von Langenbeck palatoplasty with intravelar veloplasty or the Furlow double opposing z-plasty palatoplasty between 9 and 12 months of age or between 15 and 18 months of age. Lip repair will be randomized to either the Spina or Millard method and will be accomplished by six months prior to palatoplasty. The major emphasis will focus on assessment of the near and long term outcomes of the palatal surgeries on velopharyngeal function for speech.

ELIGIBILITY:
Inclusion Criteria:

* Unrepaired unilateral cleft lip and palate
* Lip repair surgery to be accomplished by 3-6 months of age
* Able to return to research site at least once a year for follow-up

Exclusion Criteria:

* Patients with concomitant conditions (ie. mental retardation, deafness)
* Patients with Simonart Band of the cleft
* Patients who could not return to research site on a yearly basis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 1996-02; Primary Completion 2006-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Velopharyngeal function for speech was identified to be better for patients who received the Furlow double opposing z-palatoplasty procedure than patients who received the von Langenbeck procedure, as determined by the Cul-de-Sac Test of Hypernasality. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William N Williams, Ph.D, Principal Investigator — Univerisity of Florida
Locations (2):
- University of Florida, Gainesville, Florida, United States
- Hospital for Rehabilitation of Craniofacial Anomalies (USP-HRAC), Bauru, São Paulo, Brazil